CLINICAL TRIAL: NCT02342405
Title: Effect of High Inspiratory Oxygen Fraction on Endothelial Function in Healthy Volunteers: a Randomized Controlled Cross-over Trial
Brief Title: High Inspiratory Oxygen Fraction on Endothelial Function in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Ismail Gögenur, Professor., Zealand University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SJ-409
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Endothelial Dysfunction
Keywords: Oxidative stress; Nitrogen oxide; Reactive oxygen species
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30% oxygen (Placebo Comparator): Inhalation of 30% oxygen
  Interventions: Other: 30% oxygen
- 80% oxygen (Experimental): Inhalation of 80% oxygen
  Interventions: Other: 80% oxygen

INTERVENTIONS:
Other: 80% oxygen
  Arms: 80% oxygen
Other: 30% oxygen
  Arms: 30% oxygen

SUMMARY:
The frequency of preoperative cardiac ischemia and the 30-days postoperative mortality is much higher than previously assumed, with approximately 10 % of patients undergoing non-cardiac surgery suffering from postoperative myocardial injury. A recent danish study furthermore showed that patients treated with a high inspiratory oxygen fraction during surgery had a higher 1 year mortality compared with patients treated with a low inspiratory fraction. This was especially significant among patients undergoing cancer surgery. A possible explanation, is that a high oxygen fraction results in oxidative stress and endothelial dysfunction.

With this randomized cross-over study we wish to investigate the effect of a high inspiratory oxygen fraction on the endothelial function among healthy male volunteers. The primary outcome is the endothelial function assessed by the EndoPat system. Secondary outcomes are changes in oxidative biomarkers. Heart rate variability (HRV) recordings will serve as a measure for the effect of oxygen on the autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 and 30 years who has given an oral and written informed consent

Exclusion Criteria:

* Smoking, or ex-smoker Any kind of medication on a daily basis History of atopic dermatitis Known familiar hypercholesterolemia History of arteriosclerotic disease in the first and second-degree relatives Known or unknown arrhythmias, as measured by the baseline HRV-recording

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction assessed by the EndoPat-system | After 2 hours of preoxygenation
  Changes in baseline pulse-wave-amplitude (PWA) after ischemia-reperfusion from the baseline PWA measurement until 5 minutes after ischemia as a measure of altered endothelial cell function caused by high inspiratory oxygen fractions

SECONDARY OUTCOMES:
Heart rate variability (HRV) after ischemia-reperfusion as a measure of altered balance in the Autonomic nervous system | Baseline measure conducted from baseline until 20 minutes of pre oxygenation. Secondary measures is conducted 20 minutes before withdrawal of the oxygen
Plasma-Malondialdehyde (MDA) | Meaured at baseline, after 2 hours of oxygenation and after 30, 60, 120, 240 minutes after the EndoPat measure
Plasma-Arginine/Asymmetric dimethylarginine(ADMA) | Meaured at baseline, after 2 hours of oxygenation and after 30, 60, 120, 240 minutes after the EndoPat measure
Plasma-Tetrahydrobiopterin | Meaured at baseline, after 2 hours of oxygenation and after 30, 60, 120, 240 minutes after the EndoPat measure
Plasma-Advanced oxidation protein products (AOPP) | Meaured at baseline, after 2 hours of oxygenation and after 30, 60, 120, 240 minutes after the EndoPat measure
Plasma-Ascorbate/Dehydroascorbate (AA/DHA) | Meaured at baseline, after 2 hours of oxygenation and after 30, 60, 120, 240 minutes after the EndoPat measure

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, MD, DMSc, Principal Investigator — Department of surgery, Køge University Hospital
Locations (1):
- UHKoge, Køge, Denmark

REFERENCES:
- [Derived] Larsen MHH, Ekeloef S, Kokotovic D, Schou-Pedersen AM, Lykkesfeldt J, Gogenur I. Effect of High Inspiratory Oxygen Fraction on Endothelial Function in Healthy Volunteers: A Randomized Controlled Crossover Pilot Study. Anesth Analg. 2017 Nov;125(5):1793-1796. doi: 10.1213/ANE.0000000000002357. PMID 28922226